CLINICAL TRIAL: NCT04077489
Title: To Observe and Determine Macular Thickness Changes Before and After Cataract Surgery
Brief Title: Effects of 23-gauge Lensecotomy Combined With Anterior Vitrectomy on Macular in Children With Congenital Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: yin ying zhao (Other)
Responsible Party: Sponsor-Investigator, yin ying zhao, Yin Ying Zhao, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WZM2016WDD
Record Dates: First submitted 2019-08-03; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Macular; Congenital Cataract
Keywords: macular thickness
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MT (Other): Macular thickness
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — To measure the MT in congenital cataracts before and after the cataract extraction with IOL implantation surgery

SUMMARY:
Congenital cataract is the main cause of form deprivation amblyopia in children. Current studies confirm that form deprivation amblyopia affects the macular development. However, there are different opinions about the effect of amblyopia on the macular thickness . Investigators have performed "cataract extraction with IOL implantation" on children with bilateral and unilateral congenital cataract. Investigators used OCT biometry to measure children's the macular thickness before and after surgery..Average sectional total thickness was automatically determined by the instrument's software using a modified Early Treatment Diabetic Retinopathy Study (ETDRS) circle grid (fovea, inner ring, and outer ring: 1 mm, 3 mm, and 6 mm. Investigators dynamically observed changes in macular to explore the retinal mechanism of form deprivation amblyopia and help guide the clinical correct understanding of postoperative follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* congenital cataract

Exclusion Criteria:

-incooperative to complete the preoperative and postoperative examinations.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-11 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
macular thickness | 6 months
  macular thickness changes before and after cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- TianTong, Beijing, China